CLINICAL TRIAL: NCT06549842
Title: Safe and Fast Radial Hemostasis Using Synergistic Strategies: SAFE & FAST Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital of Scranton (Other)
Responsible Party: Principal Investigator, Nishant Sethi, Interventional Cardiologist, Regional Hospital of Scranton
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1378751
Record Dates: First submitted 2024-08-06; First posted 2024-08-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Cardiovascular Diseases; Bleeding; Arterial Puncture; Catheter Complications; Occlusion of Artery
Keywords: Radial artery occlusion; Rebound Bleeding; Transradial access; Coronary angiography
MeSH Terms: conditions — Cardiovascular Diseases; Hemorrhage; Arterial Occlusive Diseases | interventions — Heparin

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1-Regular dose heparin (Active Comparator): Patients in this arm will be labeled as Group 1. Patients will receive a standard heparin dose (50U/Kg) with a total compression time of 2 hours using the TR band ®.
  Interventions: Drug: Heparin; Device: Terumo Radial Band
- Group 2-Low dose heparin (Experimental): Patients in this arm will be labeled as Group 2. Patients will receive a reduced heparin dose (25 U/Kg) and a compression time of 60 minutes using the VASOBand™, with simultaneous ipsilateral ulnar artery compression.
  Interventions: Drug: Heparin; Device: Vaosband

INTERVENTIONS:
Drug: Heparin — The intervention for this study is the dose of heparin. Patients randomized to group 1 will receive a heparin dose of 50U/kg and those in group 2 will receive a lower dose of heparin at 25U/kg. Recovery period for group 1 would be 2 hours whereas for group 2 would be 1 hour.
Device: Terumo Radial Band — Group 1 will receive TR band post cardiac catheterization for radial hemostasis.
  Other Names: TR Band; Radial artery compression device
  Arms: Group 1-Regular dose heparin
Device: Vaosband — Group 2 will receive Vasoband post cardiac catheterization for radial hemostasis.
  Arms: Group 2-Low dose heparin

SUMMARY:
The Safe and Fast Radial Hemostasis using Synergistic Strategies (SAFE & FAST) trial is an interventional study aimed at reducing the incidence of radial artery occlusion (RAO) rebound bleeding, and the required compression time after transradial approach (TRA) procedures, which have become the default access for coronary procedures globally. The hypothesis is that combining lower-dose heparin and radial hemostasis with simultaneous ipsilateral ulnar artery compression could achieve these improved outcomes.

DETAILED DESCRIPTION:
Patients referred for diagnostic trans-radial cardiac catheterization who meet the inclusion criteria will be randomized into two groups. Group 1 will receive a standard heparin dose (50 U/Kg) with a total compression time of 2 hours using the TR band ® . Group 2 will receive a reduced heparin dose (25 U/Kg) and a compression time of 60 minutes using the VASOBand™, with simultaneous ipsilateral ulnar artery compression.

The study's primary endpoint is a composite of rebound bleeding, post-procedural RAO, and hematoma formation. Radial artery patency will be evaluated using ultrasonography.

With an expected complication rate of 8.2% in Group 1 and 4.5% in Group 2, a sample size of 207 patients per group will provide an 80% power to demonstrate non-inferiority for the treatment group at the alpha 2.5% level. The statistical analysis plan will use descriptive statistics for baseline data and 95% confidence intervals for outcome variables. If non-inferiority is demonstrated, there will be a superiority test performed to examine if Group 2 is superior.

In conclusion, the SAFE & FAST trial intends to establish a safer, quicker protocol for hemostasis after TRA procedures, with the potential to reduce patient recovery time and improve procedure throughput in cardiac catheterization laboratories.

ELIGIBILITY:
Inclusion Criteria:

1. Patients referred for diagnostic transradial cardiac catheterization
2. Age ≥ 18 years
3. Ability to provide written informed consent

Exclusion Criteria:

1. Absence of written informed consent
2. Patients on long-term systemic anticoagulation therapy for a different indication
3. Patients requiring a heparin dose of greater than 50 units per kilogram before, during, or after the procedure for any reason.
4. Patients requiring greater than 6 French catheter access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-08-15 (Actual); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Rebound bleeding | 24 hours
  Rebound bleeding necessitating the reapplication of the hemostatic compression.
Radial artery occlusion | 24 hours
  Post-procedural predischarge radial artery occlusion is evaluated between 30 minutes and 24 hours after the procedure.
Hematoma formation | 24 hours
  Hematoma formation during or after the procedure as ranked by the EASY criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Nishant Sethi, MD, Principal Investigator — Regional Hospital of Scranton
Locations (2):
- Regional Hospital of Scranton, Scranton, Pennsylvania, United States
- Apex Heart Institute, Ahmedabad, Gujarat, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Radial Artery Occlusion After Transradial Interventions: A Systematic Review and Meta-Analysis — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4859386/
- See also: Influence of the ratio between radial artery inner diameter and sheath outer diameter on radial artery flow after transradial coronary intervention — http://onlinelibrary.wiley.com/doi/10.1002/(SICI)1522-726X(199902)46:2%3C173::AID-CCD12%3E3.0.CO;2-4
- See also: Efficacy and safety of transient ulnar artery compression to recanalize acute radial artery occlusion after transradial catheterization — http://www.ajconline.org/article/S0002-9149(11)00469-3/abstract
- See also: Multicenter Randomized Evaluation of High Versus Standard Heparin Dose on Incident Radial Arterial Occlusion After Transradial Coronary Angiography: The SPIRIT OF ARTEMIS Study — https://pubmed.ncbi.nlm.nih.gov/30391389/
- See also: Randomized Trial of Compression Duration After Transradial Cardiac Catheterization and Intervention — http://www.ahajournals.org/doi/full/10.1161/JAHA.116.005029?rfr_dat=cr_pub++0pubmed&url_ver=Z39.88-2003&rfr_id=ori%3Arid%3Acrossref.org
- See also: Randomized clinical trial on short-time compression with Kaolin-filled pad: a new strategy to avoid early bleeding and subacute radial artery occlusion after percutaneous coronary intervention — http://pubmed.ncbi.nlm.nih.gov/20807305/
- See also: The Leipzig prospective vascular ultrasound registry in radial artery catheterization: impact of sheath size on vascular complications — https://pubmed.ncbi.nlm.nih.gov/22230148/
- See also: Interruption of blood flow during compression and radial artery occlusion after transradial catheterization — http://onlinelibrary.wiley.com/doi/10.1002/ccd.21058
- See also: Incidence, predictors, and clinical impact of bleeding after transradial coronary stenting and maximal antiplatelet therapy — https://www.proquest.com/docview/1504614575?sourcetype=Scholarly%20Journals
- See also: Randomized COmparison of Isolated Radial Artery ComPrEssioN Versus Radial and Ipsilateral Ulnar Artery Compression in Achieving Radial Artery Patency: The OPEN-Radial Trial — http://pubmed.ncbi.nlm.nih.gov/32961529/